CLINICAL TRIAL: NCT03381170
Title: An Open Label Extension of the TG1101-RMS201 Trial, for Subjects Currently Enrolled in TG1101-RMS201Treated With Ublituximab for Relapsing Forms of Multiple Sclerosis
Brief Title: An Extension of the TG1101-RMS201 Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TG1101-RMS201E
Record Dates: First submitted 2017-12-18; First posted 2017-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Relapsing Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — ublituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ublituximab (Experimental): Ublituximab IV infusions on Weeks 1E, 24E, 48E, 72E and (6E
  Interventions: Biological: Ublituximab

INTERVENTIONS:
Biological: Ublituximab — Enrolled Subjects will be infused with ublituximab on Weeks 1E, 24E, 48E, 72E and 96E
  Other Names: TG1101

SUMMARY:
This study evaluates the long term use of a single agent ublituximab, a novel monoclonal antibody, in patients with relapsing forms of multiple sclerosis

ELIGIBILITY:
Inclusion Criteria:

* Subjects currently enrolled in TG1101-RMS201 trial
* Subjects who have completed three infusions of ublituximab (at Day 1, Day 15, and Week24, as specified in the TG1101-RMS201 protocol) and have completed the scheduled assessments up to the final 48-week visit

Exclusion Criteria:

* Subjects who discontinued ublituximab treatment or withdrew consent from the TG1101- RMS201 study during the 48-week evaluation period
* Subjects who have started any other immunomodulating or disease modifying therapy after completion of the TG1101-RMS201 trial
* Pregnant or nursing mothers

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related events as assessed by CTCAE V4.0 | 96 weeks on therapy
  to determine the incidence of adverse events and any abnormal laboratory values

SECONDARY OUTCOMES:
Evaluate the % of participants with relapses | up to 96 Weeks

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - TG Therapeutics Investigational Trial Site, Pasadena, California
  - TG Therapeutics Investigational Trial Site, Aurora, Colorado
  - TG Therapeutics Investigational Trial Site, Lexington, Kentucky
  - TG Therapeutics Investigational Trial Site, Columbus, Ohio
  - TG Therapeutics Investigational Trial Site, Westerville, Ohio
  - TG Therapeutics Investigational Trial Site, Knoxville, Tennessee
  - TG Therapeutics Investigational Trial Site, Round Rock, Texas
  - TG Therapeutics Investigational Trial Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared after study completion via publication